CLINICAL TRIAL: NCT05545449
Title: Barriers to Adolescent PrEP in Western Kenya: An Implementation Sciences Approach
Brief Title: Adapting an Adolescent Friendly PrEP Program for Uasin Gishu County-Kenya
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Academic Model Providing Access to Healthcare (AMPATH) (Other); Indiana CTSI (Unknown)
Responsible Party: Principal Investigator, Mary A. Ott, Professor of Pediatrics, Indiana University
Other Study IDs: IUIRB-13771
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV Pre-exposure Prophylaxis; Stigma, Social
Keywords: Peer mentor; Global health; Adolescent
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: PrEP Peer Mentor Program — Five PrEP peer mentors will provide outreach, education, and referral for HIV pre-exposure prophylaxis. Peer mentors have received training on HIV, PrEP, family planning, adolescent development, peer support, and action planning. Interactions will include 1:1 informal interactions as well as planned group outreach interactions.

SUMMARY:
The purpose of this study is to examine the implementation ( e.g. training, reach, acceptability) of a a youth friendly pre-exposure prophylaxis (PrEP) peer mentorship program for Adolescents and Young Adults (AYA). This program will include the use of PrEP focused peer-mentors for education on HIV risk and on PrEP as well as for support for those who end up starting PrEP. This will be an adaptation from the HIV peer mentor program which has been successfully utilized at the Academic Model Providing Access to Healthcare (AMPATH) to improve on the outcomes of Adolescents Living with HIV. Investigators use the Exploration, Preparation, Implementation and Sustainment (EPIS) implementation science framework to guide our research process and address our implementation aims. We will use both qualitative (key stakeholder focus group discussions (FGDs)) and quantitative data collection methods (electronic health records (EHR) review) to evaluate the acceptability and change in knowledge and number of adolescents.

DETAILED DESCRIPTION:
This study pilots the implementation of an intervention (AYA PrEP peer mentors) in increasing knowledge, reducing stigma and increasing uptake and adherence to PrEP among AYA. In low and middle income countries, peer mentor interventions to improve health behaviors are well supported by evidence, and used extensively by the AMPATH programs as a best practice. We are examining the implementation (e.g. training, reach, acceptability) rather than the effectiveness of this intervention. The study has been approved by both the IU IRB and the Moi University Institutional Research Ethics Committee.

The intervention will engage five PrEP focused peer-mentors, one stationed at Moi Teaching and Referral Hospital Reproductive Health Clinic; one from the Lesbian, Gay, Bisexual, Transgender, and Queer (LGBTQ) community, and three from specified tertiary institutions in Eldoret, Kenya (Eldoret Medical Training College, The University of Eldoret, Eldoret Polytechnic) to focus on college students. These peer mentors will be paid a monthly stipend, and their roles will be to: (1) Hold one on one discussions with target AYA on PrEP; (2) To hold group discussions on PrEP with the target AYA; (3) To champion for PrEP promotion and provision by healthcare workers; and (4) To do outreach-work, adherence support and clinic reminders for those on PrEP. Peer mentors received PrEP and peer mentor training adapted from an existing USAID curriculum, as well as training in research procedures. Peer mentors will complete a pre-and post-training survey to measure their efficacy and knowledge on HIV and PrEP.

The EHR aspect of the study will involve extraction of data before and during the peer mentor intervention. The data extraction will include de-identified information from visits for PrEP initiation and PrEP maintenance among AYA in Uasin Gishu County. We will collect the socio-demographic and clinical data of PrEP initiation and maintenance visits among AYA aged 15-24 years. The qualitative data aspects will involve FGDs with 1) the PrEP focused peer mentors, 2) PrEP AYA initiators, and 3) Healthcare workers. This FGDs will explore the acceptability, feasibility and adaption of the AYA PrEP peer mentor program. The quantitative data will also include PrEP peer mentors completing a tracking form that describes characteristics of the outreach interaction, including the total # people, topics discussed, and whether the group was a high risk group (e.g. LGBTQ, pregnant/parenting, discordant relationship). No personal identifiers or identifiable characteristics of individuals will be collected, and a waiver of informed consent has been granted.

For data analysis to look at effectiveness, the number of visits for PrEP initiation and maintenance in the system for a 3 month period before the intervention starts will be compared to the number of visits for PrEP initiation during the intervention. De-identified EHR data will be used. To qualitatively examine the effect of the intervention on stigma and barriers, FGDs will be conducted with AYA, healthcare workers, and peer mentors at the end of the intervention. To examine the implementation of the intervention, (1) the number of of participants overall, (2) the total number of interactions/outreach, (3) the total number of interactions/outreach that include someone from higher HIV risk groups, and (4) the topics of the outreach interaction will be tracked using run charts.

ELIGIBILITY:
Inclusion Criteria:

* for FGD: 18-24 year old AYAs, peer mentors, and health care providers.
* for EHR: 15-24 year olds initiating and maintaining PrEP
* from peer mentor tracking: 15-24 year old interacting with peer mentors

Exclusion Criteria:

* for FGD: unable to speak English or Swahili, intoxicated or high

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * For Focus Group Discussions: (1) 18-24 year olds AYA selected from PrEP users identified from the EMR (n=12); (2) peer mentors (all 5); (3) health care staff/providers (n=12).
  * For EMR review: 15-24 year olds attending AMPATH clinics in Uasin Gishu county for PrEP initiation or maintenance.
  * For peer mentor tracking: 15-24 year olds interacting with peer mentors.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
AYA EHR visits for PrEP initiation and maintenance. | 3 months before and the 1 year duration of the intervention
  The number of visits for PrEP initiation and maintenance in the AMPATH EHR system.

SECONDARY OUTCOMES:
Number of AYA reached by PrEP peer mentors | Monthly for 1 year
  For each peer mentor interaction (both informal discussions and formal group outreach), peer mentors will complete a tracking that captures number of individuals in the outreach/interaction.
Number and proportion of peer mentor interactions involving individuals from higher risk group | Monthly for 1 year
  For each interaction (both informal discussions and formal group outreach), peer mentors will complete a tracking that captures number of individuals in the outreach/interaction, the age range, and whether the interaction/outreach included anyone from a high risk group (e.g. LGBTQ, pregnant, serodiscordant). We will examine the total number of interactions (both formal and information) and the number and proportion involving a higher risk group.
Number of peer mentor interactions resulting in referrals for PrEP | Monthly for 1 year
  The Peer Mentor tracking forms collect whether anyone in the outreach/interaction is referred for PrEP. We will identify the number of interactions resulting referrals resulting from PrEP peer mentor outreach interactions.

OTHER OUTCOMES:
PrEP stigma | Focus groups will be conducted 9-12 months after the start of the intervention
  From focus group discussions we will describe participants' perceptions of PrEP stigma expressed by peer mentors, AYA, and health care providers, including the type of stigma and the effects of stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Ott, MD MA, Principal Investigator — Icahn School of Medicine at Mount Sinai; Juddy Wachira, PhD, Principal Investigator — Moi University; Edith Apondi, MBChB MMed, Principal Investigator — Academic Model Providing Access to Healthcare
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Undecided
A data package including focus group transcripts, EHR data, and peer mentor tracking forms will be created.